CLINICAL TRIAL: NCT03740438
Title: Modeling of the Hemoglobin Drop in the Uncomplicated Postoperative Course
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Sebastian Jaramillo, Principal Investigator, Hospital Clinic of Barcelona
Other Study IDs: HCB/2016/0906/2
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Surgical Blood Loss; Surgery; Perioperative/Postoperative Complications
Keywords: Hemoglobin; Hemoglobin drop; Surgical Blood loss
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Complications | interventions — Erythrocyte Indices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hemoglobin concentration — Perioperative hemogloin concentration

SUMMARY:
transfusion-related decisions in the perioperative setting are often complex due to acute variations in the hemoglobin levels, which typically experience a progressive decrease within days. This process, commonly referred to as "hemoglobin drop" or "hemoglobin drift", has been observed to be highly variable among patients and reliant on several variables, such as the volemic status, fluid balance and blood loss. Although it has been investigated and some predictors have been identified, postoperative hemoglobin drop remains unpredictable and is not fully clarified. In consequence, hemoglobin levels' variations are frequently misunderstood, hindering the decision to transfuse.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients electively scheduled for laparoscopic urologic and gynecologic surgery.

Exclusion Criteria:

* Suspected or confirmed coagulopathy (including current treatment with anticoagulants or antiplatelet agents).
* Requirement for surgical gauzes during surgery, including conversion to open surgical techniques.
* Transfusion of red blood cells (RBCs) or use of blood recovery systems during the perioperative period.
* Significant postoperative bleeding (> 50 ml in surgical drains, gross hematuria, or any other type of significant blood loss).
* Postoperative hemodynamic instability (defined as requirement of vasoactive drugs).
* Other major postoperative complications during the observable period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients electively scheduled for laparoscopic urologic and gynecologic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration | 2-5 days
  Patient´s hemoglobin concentration in the postoperative course (measured every 24 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided